CLINICAL TRIAL: NCT03080142
Title: Transversus Abdominus Plane (TAP) Block Catheters vs Liposomal Bupivacaine for Pain Control After Colorectal Surgery: A Prospective Randomized Control Trial
Brief Title: TAP Block Catheters vs Liposomal Bupivacaine for Pain Control After Colorectal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 983837
Record Dates: First submitted 2017-03-09; First posted 2017-03-15 (Actual); Results first posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Colorectal Surgery; TAP Blocks
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Single injection of Exparel
  Interventions: Drug: Exparel
- Group 2 (Active Comparator): Injection of Ropivicaine (Naropin) bolus and placement of Ropivicaine catheters
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Exparel — Patients will receive an injection of 30ml of volume to each abdominal side with a total of 60 ml for bilateral TAP blocks.
  Other Names: Bupivacaine liposome injectable suspension
  Arms: Group 1
Drug: Ropivacaine — Patients will receive 30ml of ropivicaine. Peripheral nerve catheters will be placed approximately 3-5cm into the TAP space and secured to the skin with tegaderm tape. Infusions will be ordered with CADD pumps and will be initiated at a rate of 8ml/hr of 0.2% ropivicaine on the inpatient floor.
  Other Names: Naropin
  Arms: Group 2

SUMMARY:
This is a prospective randomized study designed to compare the pain control from a single shot of liposomal bupivacaine (Exparel) against transversus abominus plane (TAP) catheters with ropivicaine bolus in patients undergoing elective colorectal surgery.

DETAILED DESCRIPTION:
At UC Davis, it is standard practice to place TAP blocks with catheters for adult colorectal surgery patients for perioperative pain control. This practice, however, is resource intensive, adds the risk of catheter-related complications, and adds increased burden to patients by requiring them to be tethered to 2 catheters.

An alternative TAP can be performed using a single shot of liposomal bupivacaine (Exparel), an extended release local anesthetic that is FDA-approved for surgical plane infiltration including TAP blocks.

With this prospective study, we seek to improve patient care at UC Davis and educate other institutions through the use of concrete data comparing these 2 treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective colorectal surgery with Dr. Linda Farkas

Exclusion Criteria:

* Patients under 18 years of age
* Patient over 90 years of age
* Pregnancy
* Prisoners
* Patients unable to provide consent
* Patients on systemic anticoagulation therapy
* Patients with an allergy to local anesthetics

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Zhou, MD, Principal Investigator — UC Davis Health
Locations (1):
- UC Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Liposomal Bupivacaine Group: Single injection of Exparel
  Exparel: Patients will receive an injection of 30ml of volume to each abdominal side with a total of 60 ml for bilateral TAP blocks.
- Ropivacaine Catheter Group: Injection of Ropivicaine (Naropin) bolus and placement of Ropivicaine catheters
  Ropivacaine: Patients will receive 30ml of ropivicaine. Peripheral nerve catheters will be placed approximately 3-5cm into the TAP space and secured to the skin with tegaderm tape. Infusions will be ordered with CADD pumps and will be initiated at a rate of 8ml/hr of 0.2% ropivicaine on the inpatient floor.
Period: Overall Study
Arm/Group | Liposomal Bupivacaine Group | Ropivacaine Catheter Group
Started | 42 | 44
Completed | 42 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 42 | 44 | 86
Age, Continuous [Mean (Full Range); unit: years] | 57.4 [19 to 79] | 57.1 [19 to 80] | 57.2 [19 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 45
  Male | 21 | 20 | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 42 | 44 | 86

OUTCOME MEASURES:

1. Primary Outcome: Mean Opioid Consumption in Morphine Opioid Equivalents in mg
Description: Anticipate superior efficacy and pain control with liposomal bupivacaine TAP blocks measured by use of opioids (measured in oral morphine equivalents) in the first 48 hours following surgery
  Will use opioid consumption in morphine equivalents as a comparison
Time Frame: 48 hours from start of surgery
Measure: Mean (Standard Deviation); unit: IV morphine equivalents (mg)
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 42 | 44
IV morphine equivalents (mg) | 112.12 (112.8) | 97.95 (58.15)

ADVERSE EVENTS:
Time Frame: From study enrollment in the preoperative holding area for 2 hospital days
Description: No adverse events with patients enrolled in this study
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/44
Other Adverse Events (participants affected / at risk) | 0/42 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT03080142/Prot_SAP_001.pdf
  • Informed Consent Form (2017-03-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT03080142/ICF_000.pdf